CLINICAL TRIAL: NCT03272724
Title: French National Observatory on Infective Endocarditis
Acronym: ObservatoireEI
Status: Recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Bichat Hospital (Other); Centre Hospitalier Universitaire de la Guadeloupe (Other); Centre Hospitalier Universitaire de Besancon (Other); Hospices Civils de Lyon (Other); University Hospital, Montpellier (Other); Rennes University Hospital (Other); Hôpital Saint André, Reims (Unknown); Henri Mondor University Hospital (Other); Polyclinique Courlancy, Reims (Unknown); Centre Hospitalier Universitaire de Saint Etienne (Other); Bicetre Hospital (Other); Centre Hospitalier Universitaire, Amiens (Other); Centre Hospitalier Universitaire Dijon (Other); Centre Hospitalier Annecy Genevois (Other); Centre Hospitalier de Roanne (Other); Centre hospitalier Pierre Oudot Bourgoin-Jallieu (Unknown); L'hôpital Nord-Ouest - Villefranche Villefranche sur Saône (Other); Hôpital d'Instruction des Armées Desgenettes (Other); Hôpital intercommunal Sud Léman Valserine, Saint Julien en Genevois (Unknown); University Hospital, Grenoble (Other); Centre Cardiologique du Nord (Other); Centre Hospitalier Intercommunal Robert Ballanger (Other); Raincy Montfermeil Hospital Group (Network); Pitié-Salpêtrière Hospital (Other); Hôpital Cochin (Other); Hospital Avicenne (Other); Beaujon Hospital (Other); European Georges Pompidou Hospital (Other); Hopital Foch (Other); Hotel Dieu Hospital (Other); Hôpital Jean Verdier (Other); Hopital Lariboisière (Other); Hôpital Necker-Enfants Malades (Other); Fondation Hôpital Saint-Joseph (Other); Saint-Louis Hospital, Paris, France (Other); Tenon Hospital, Paris (Other); Saint Antoine University Hospital (Other); Centre hospitalier de Saint Dié des Vosges (Unknown); Centre Hospitalier Régional Metz-Thionville (Other); Hôpital d'Instruction des Armées Legouest (Other); Hôpital sainte Blandine Metz (Unknown); Hôpital-clinique Claude Bernard, Metz (Unknown); Polyclinique Louis Pasteur Essey-les-Nancy (Unknown); Hopital Nord Franche-Comte (Other); Lons le Saunier hospital (Unknown); Pontarlier hospital (Unknown); Epernay hospital (Unknown); Chalons en Champagne hospital (Unknown); Clinique Saint Vincent Epernay (Unknown); Hôpital Maison Blanche Reims (Unknown); Hopital Universitaire Robert-Debre (Other); Beziers Hospital (Other); Louis Pasteur hospital, Bagnols sur Cèze (Unknown); Centre hospitalier de Perpignan (Other); Narbonne Hospital (Other); Clinique du Millenaire (Other); Centre Hospitalier Universitaire de Nīmes (Other); Saint Malo hospital (Unknown); HIA Begin, Saint Mandé (Unknown); Centre Hospitalier d'Alès-Cévennes (Unknown); University Hospital, Bordeaux (Other); Centre hospitalier de Chambéry (Unknown); Poitiers University Hospital (Other); Centre Hospitalier Intercommunal Villeneuve Saint Georges (Unknown); Centre Hospitalier Argenteuil (Other); Hospital St. Joseph, Marseille, France (Other); Centre hospitalier de Vannes (Unknown); University Hospital, Strasbourg, France (Other); Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Principal Investigator, Christine Selton-Suty, Dr, Central Hospital, Nancy, France
Other Study IDs: Observatoire EI
Record Dates: First submitted 2017-08-28; First posted 2017-09-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this observatory is to provide a national database of infective endocarditis, informed by all volunteer centers, using a standardized case report forms.

Such an observatory will describe the clinical profile, microbiological, therapeutic and evolving of infective endocarditis (IE); analyze the risk factors for the disease and its prognosis factors of evolution; describe management practices; evaluate and compare in the real drug treatment strategies (including antibiotics) and surgical.

DETAILED DESCRIPTION:
All the clinical, biological, microbiological and laboratory describing the history of patients and their evolution during hospitalization for infective endocarditis will be obtained from physicians supporting patients and recorded in an electronic case report form. Will include collected clinical characteristics (site, pre-existing heart disease underlying symptoms, complications), biological characteristics (dosage on admission and diagnosis), microbiological characteristics (identifying the genus and species of the microorganism responsible, sensitivity to antibiotics susceptibility testing and evaluated by determination of minimal inhibiting concentration (MIC), exhaustive search of the rare forms of endocarditis uncultivated microorganisms), an analysis of the gateways based on the causative organism; echocardiographic characteristics (number and size of vegetations, valvular damage, scalable: surgery, lethality) and therapeutic characteristics (antibiotic treatment, surgical).

ELIGIBILITY:
Inclusion Criteria:

* Major Patient
* Supported in one of the participating centers
* The application of diagnostic classification criteria of Duke modified by Li is carried out after collection of all the data at the end of the patient's hospitalization. Only patients meeting criteria for definite or possible endocarditis will be included in the analyses.
* Registered with the French social security system

Exclusion Criteria:

• Refusal of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients, suspected of infective endocarditis
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 1991-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
history of heart disease | inclusion
  status of heart valves, pre-existing heart conditions
risk factors, medical history | inclusion
  associated diseases
origin of infection | period of 3 months before infective endocarditis
  high risk procedures
weight | inclusion
  kg
height | inclusion
  cm
clinical symptoms | inclusion
  cardiac, peripheral and neurological symptoms
biological outcomes | inclusion
  blood count
microbiological outcomes | inclusion
  identification of infecting organisms
diagnostic imaging | inclusion
  description of tyhe imaging tests performed
antibiotic therapy | from inclusion to recovery
  antibiotic treatment: type and duration
surgical procedures | from inclusion to recovery
  description of surgical procedures

SECONDARY OUTCOMES:
biologic collection (optional) | inclusion
  plasma and serum collection

CONTACTS AND LOCATIONS:
Overall Officials: Christine SELTON-SUTY, MD, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lefevre B, Habib G, Hoen B, Selton-Suty C, Philip M, Issa N, Danneels P, De La Chapelle M, Deschanvres C, Erpelding ML, Tattevin P, Le Bot A, Villamarin M, Fernandez-Hidalgo N, Tribouilloy C, Pluquet E, Dubee V, Hannan M, Dornikova G, Durante-Mangoni E, Bertolino L, Siciliano RF, Amaral de Oliveira AM, Goulart Correia M, Gouriet F, Lamas C. Staphylococcus lugdunensis infective endocarditis: a multicentre international observational study. Infect Dis (Lond). 2025 Sep 15:1-9. doi: 10.1080/23744235.2025.2556921. Online ahead of print. PMID 40952378
- [Background] Selton-Suty C, Goehringer F, Venner C, Thivilier C, Huttin O, Hoen B; membres de l'Endocarditis Team du CHU de Nancy. [Complications and prognosis of infective endocarditis]. Presse Med. 2019 May;48(5):532-538. doi: 10.1016/j.lpm.2019.04.002. Epub 2019 May 2. French. PMID 31056233
- [Background] Hoen B, Elfarra M, Huttin O, Goehringer F, Venner C, Selton-Suty C; l'Endocarditis Team du CHU de Nancy. [Treatment of infectious endocarditis]. Presse Med. 2019 May;48(5):539-548. doi: 10.1016/j.lpm.2019.04.015. Epub 2019 May 18. French. PMID 31109766
- [Background] N'Guyen Y, Duval X, Revest M, Saada M, Erpelding ML, Selton-Suty C, Bouchiat C, Delahaye F, Chirouze C, Alla F, Strady C, Hoen B; AEPEI study group. Time interval between infective endocarditis first symptoms and diagnosis: relationship to infective endocarditis characteristics, microorganisms and prognosis. Ann Med. 2017 Mar;49(2):117-125. doi: 10.1080/07853890.2016.1235282. Epub 2016 Nov 3. PMID 27607562
- [Background] Lefevre B, Hoen B, Goehringer F, Sime WN, Aissa N, Alauzet C, Jeanmaire E, Henard S, Filippetti L, Selton-Suty C, Agrinier N; for AEPEI study group (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse). Antistaphylococcal penicillins vs. cefazolin in the treatment of methicillin-susceptible Staphylococcus aureus infective endocarditis: a quasi-experimental monocentre study. Eur J Clin Microbiol Infect Dis. 2021 Dec;40(12):2605-2616. doi: 10.1007/s10096-021-04313-3. Epub 2021 Aug 12. PMID 34383175
- [Background] Collonnaz M, Erpelding ML, Alla F, Goehringer F, Delahaye F, Iung B, Le Moing V, Hoen B, Selton-Suty C, Agrinier N; AEPEI Study Group. Impact of referral bias on prognostic studies outcomes: insights from a population-based cohort study on infective endocarditis. Ann Epidemiol. 2021 Feb;54:29-37. doi: 10.1016/j.annepidem.2020.09.008. Epub 2020 Sep 18. PMID 32950657
- [Background] Collonnaz M, Erpelding ML, Alla F, Goehringer F, Delahaye F, Iung B, Le Moing V, Hoen B, Selton-Suty C, Agrinier N; AEPEI study group. Data on prognostic factors associated with 3-month and 1-year mortality from infective endocarditis. Data Brief. 2020 Nov 1;33:106478. doi: 10.1016/j.dib.2020.106478. eCollection 2020 Dec. PMID 33225027
- [Background] De Ciancio G, Erpelding ML, Filippetti L, Goehringer F, Blangy H, Huttin O, Agrinier N, Juilliere Y, Sadoul N, Selton-Suty C. Adherence to diagnostic and therapeutic practice guidelines for suspected cardiac implantable electronic device infections. Arch Cardiovasc Dis. 2021 Oct;114(10):634-646. doi: 10.1016/j.acvd.2021.06.010. Epub 2021 Nov 3. PMID 34742672
- [Background] Selton-Suty C, Delahaye F, Tattevin P, Federspiel C, Le Moing V, Chirouze C, Nazeyrollas P, Vernet-Garnier V, Bernard Y, Chocron S, Obadia JF, Alla F, Hoen B, Duval X; AEPEI (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse). Symptomatic and Asymptomatic Neurological Complications of Infective Endocarditis: Impact on Surgical Management and Prognosis. PLoS One. 2016 Jul 11;11(7):e0158522. doi: 10.1371/journal.pone.0158522. eCollection 2016. PMID 27400273
- [Background] Radjabaly Mandjee A, Filippetti L, Goehringer F, Duval X, Botelho-Nevers E, Tribouilloy C, Huguet R, Chirouze C, Erpelding ML, Hoen B, Selton-Suty C, Agrinier N, Lefevre B; investigators of the French AEPEI Observatory on Infective Endocarditis (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse). Characteristics of patients with infective endocarditis and no underlying cardiac conditions. Infect Dis (Lond). 2022 Sep;54(9):656-665. doi: 10.1080/23744235.2022.2078404. Epub 2022 May 23. PMID 35604065
- [Background] Beraud G, Tubiana S, Erpelding ML, Le Moing V, Chirouze C, Gorenne I, Manchon P, Tattevin P, Vernet V, Varon E, Hoen B, Duval X; AEPEI study group; COMBAT study group. Combined Bacterial Meningitis and Infective Endocarditis: When Should We Search for the Other When Either One is Diagnosed? Infect Dis Ther. 2022 Aug;11(4):1521-1540. doi: 10.1007/s40121-022-00651-7. Epub 2022 May 26. PMID 35618954
- [Background] Lefevre B, Legoff A, Boutrou M, Goehringer F, Ngueyon-Sime W, Chirouze C, Revest M, Vernet Garnier V, Duval X, Delahaye F, Le Moing V, Selton-Suty C, Filippetti L, Hoen B, Agrinier N. Staphylococcus aureus endocarditis: Identifying prognostic factors using a method derived from morbidity and mortality conferences. Front Med (Lausanne). 2022 Dec 6;9:1053278. doi: 10.3389/fmed.2022.1053278. eCollection 2022. PMID 36561723
- [Background] Fowler VG, Durack DT, Selton-Suty C, Athan E, Bayer AS, Chamis AL, Dahl A, DiBernardo L, Durante-Mangoni E, Duval X, Fortes CQ, Fosbol E, Hannan MM, Hasse B, Hoen B, Karchmer AW, Mestres CA, Petti CA, Pizzi MN, Preston SD, Roque A, Vandenesch F, van der Meer JTM, van der Vaart TW, Miro JM. The 2023 Duke-International Society for Cardiovascular Infectious Diseases Criteria for Infective Endocarditis: Updating the Modified Duke Criteria. Clin Infect Dis. 2023 Aug 22;77(4):518-526. doi: 10.1093/cid/ciad271. PMID 37138445
- [Background] El Hatimi S, Erpelding ML, Selton-Suty C, Botros JB, Goehringer F, Berthelot E, Elfarra M, Deconinck L, Para M, Provenchere S, Hoen B, Agrinier N, Duval X, Iung B. Predictive performance of surgical mortality risk scores in infective endocarditis. Eur J Cardiothorac Surg. 2024 Jan 2;65(1):ezad433. doi: 10.1093/ejcts/ezad433. PMID 38175782
- [Background] Bucy L, Erpelding ML, Boursier C, Lefevre B, Alauzet C, Liu Y, Chevalier E, Huttin O, Agrinier N, Selton-Suty C, Goehringer F; AEPEI study group (Association pour l'Etude et la Prevention de l'Endocardite Infectieuse). Real world experience of therapeutic monitoring of medically treated prosthetic valve infective endocarditis by 18F-FDG-PET/CT. J Nucl Cardiol. 2023 Oct;30(5):2096-2103. doi: 10.1007/s12350-023-03339-8. Epub 2023 Jul 31. PMID 37524996
- [Background] Goehringer F, Lalloue B, Selton-Suty C, Alla F, Botelho-Nevers E, Chirouze C, Curlier E, El Hatimi S, Gagneux-Brunon A, le Moing V, Lim P, Piroth L, Strady C, Tribouilloy C, Virion JM, Agrinier N, Duval X, Hoen B; Association pour l'Etude et la Prevention de l'Endocardite Infectieuse-ObservatoireEI Study Group. Compared Performance of the 2023 Duke-International Society for Cardiovascular Infectious Diseases, 2000 Modified Duke, and 2015 European Society of Cardiology Criteria for the Diagnosis of Infective Endocarditis in a French Multicenter Prospective Cohort. Clin Infect Dis. 2024 Apr 10;78(4):937-948. doi: 10.1093/cid/ciae035. PMID 38330171